CLINICAL TRIAL: NCT00805415
Title: Multicenter, Open-label, Randomized, Comparative Study to Evaluate Ovulation Inhibition With Two 4-phasic Oral Contraceptive Regimens Containing Estradiol Valerate and Dienogest Applied Daily for Three Cycles to 200 Healthy Female Volunteer
Brief Title: Ovulation Inhibition of Two 4-phasic Oral Contraceptive Regimens
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Therapeutic Area Head, Bayer Healthcare AG
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 91271; 307300
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Ovulation Inhibition
Keywords: Oral Contraceptive; Ovulation Inhibition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: EV/DNG (Qlaira, BAY86-5027, SH T00658K)
- Arm 2 (Experimental)
  Interventions: Drug: EV/DNG (SH T00658L)

INTERVENTIONS:
Drug: EV/DNG (Qlaira, BAY86-5027, SH T00658K) — Estradiol valerate (EV) and dienogest (DNG) in a sequential 4-phasic regimen, EV 3, 2, and 1 mg and DNG 2 and 3 mg
  Arms: Arm 1
Drug: EV/DNG (SH T00658L) — Estradiol valerate (EV) and dienogest (DNG) in a sequential 4-phasic regimen, EV 3, 2, and 1 mg and DNG 3 and 4 mg
  Arms: Arm 2

SUMMARY:
The aim of the study is to investigate the ovulation inhibition of two 4-phasic oral contraceptive regimens.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women willing to use non-hormonal methods of contraception

Exclusion Criteria:

* Women with any contraindication for oral contraceptive use, for example but not limited to: presence or history of venous or arterial thrombotic / thrombembolic events, hypertension, presence or history of severe hepatic disease

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 209 (Actual)
Dates: Start 2003-03; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with a Hoogland score of 5-6 (luteinized unruptured follicle [LUF] or ovulation) | Treatment cycles 2 and 3

SECONDARY OUTCOMES:
Proportion of subjects with a Hoogland score of 5-6 (LUF or ovulation) | Treatment cycles 2 or 3
Measurements of endometrial thickness | Treatment cycles 2 and 3
Visibility of cervical mucus | Treatment cycles 2 and 3
Ovarian activity (Hoogland score) | Posttreatment cycle (only subjects from center 2)Treatment cycles 2 and 3
Measurements of follicle size | Treatment cycles 2 and 3
Measurements of hormone levels (follicle-stimulating hormone [FSH], luteinizing hormone [LH], progesterone and estradiol) | Treatment cycles 2 and 3
Compliance | Throughout whole study
Medical, surgical and medication history, concomitant medication, general physical and gynecological examination, cervical smear, pregnancy test, adverse events, safety laboratory determinations, cycle control, vital signs | Various timepoint throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- Dinox GmbH Berlin, Berlin, State of Berlin, Germany
- Dinox B.V., Groningen, Netherlands